CLINICAL TRIAL: NCT02872246
Title: Sun Protection Factor (SPF) / UVA Protection Factor (UVAPF) Assay
Brief Title: Sun Protection Factor (SPF) / UVA Protection Factor (UVAPF) - Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18321
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF evaluation (Experimental): Subjects with good health as determined from the CRO Subject History Form (SHF) and Fitzpatrick Skin Type I, II and/or III were included for SPF testing.
  Interventions: Drug: BAY 987516; Drug: SPF 15 Control

INTERVENTIONS:
Drug: BAY 987516 — Single dose application of two (2) mg/cm² of test product. Each 50 cm² test site area requires 100 mg of a product to obtain a standard 2 mg/cm² test application.
Drug: SPF 15 Control — Single dose application of two (2) mg/cm² of test product. Each 50 cm² test site area requires 100 mg of a product to obtain a standard 2 mg/cm² test application.

SUMMARY:
Evaluation of the effectiveness of a sunscreen product by determining its Sun Protection Factor (SPF) on the skin of human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of an age of 18 to 70 years inclusive;
* Fitzpatrick Skin Type I, II and/or III for SPF testing;
* Good health as determined from the CRO Subject History Form (SHF);
* Signed and dated Informed Consent Form;
* Signed and dated Health Insurance Portability and Accountability Act (HIPAA) Form;
* An unambiguous minimal erythema dose (MED).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of water resistant SPF | 16-24 hours post exposure
  For the sunscreen Test Material, two test sites were used; one for before immersion and one for after 2 hours of water immersion. One additional test site area was used for the control SPF determination, on each subject, as per the COLIPA Sun Protection Factor Test Method.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Union, New Jersey, United States